CLINICAL TRIAL: NCT01816269
Title: Effect of Dental Scaling on Helicobacter Pylori Eradication and Reinfection
Acronym: Scaling and Hp
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Goztepe Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Celal Ulasoglu, MD Department of Gastroenterology, Goztepe Training and Research Hospital
Other Study IDs: cu1959
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Dental scaling; Eradication; Reinfection; Helicobacter status
MeSH Terms: conditions — Reinfection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with scaling and patients without scaling: No drug
- Helicobacter eradicated or non-eradicated

SUMMARY:
Patients who had received H.pylori eradication treatment will be categorised as eradication and reinfection status and whether dental scaling has any influence on these results.

DETAILED DESCRIPTION:
Patients over 18 years with no comorbidities especially liver, cardiac and haemorrhagic diathesis and giving informed consent will be categorised according to their status of dental scaling, eradication and reinfection rates of h.pylori.

Statistical examination will include the multiple regression and Chi-Square.

The result will emphasize the influence of dental scaling on eradication (Presence of Hp cure 1-6 months after treatment) and reinfection ( reappearance of Hp 12 months later than the treatment).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 with h.pylori positivity and received anti-Hp treatment giving informed consent to analyse of their data on this subject.

Exclusion Criteria:

* Comorbidities with cardiac, liver and medical contraindication to perform dental scaling.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible population with H.pylori infection and result of treatment based on presence of dental scaling.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-03; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
The eradication and reinfection rates in dental scaled and non-scaled patients. | last 1 year

SECONDARY OUTCOMES:
Reinfection rate of patients treated for H.pylori | 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - GoztepeTRH, Istanbul, Istanbul
  - GoztepeTRH, Istanbul